CLINICAL TRIAL: NCT01544283
Title: Heated Lidocaine Patch Compared to Subacromial Injections in the Treatment of Pain Associated With Shoulder Impingement Syndrome, A Pilot
Brief Title: Pain Patch Versus Injections in the Treatment of Pain Associated With Shoulder Impingement Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Injury Care Medical Center (Other)
Collaborators: Nuvo Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NS001
Record Dates: First submitted 2012-02-23; First posted 2012-03-05 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Shoulder Pain
Keywords: Shoulder Pain; Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Pain; Shoulder Impingement Syndrome | interventions — Lidocaine; Tetracaine; Transdermal Patch; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patch (Experimental): Patch will be applied directly to the lateral tip of the affected shoulder, at the site of maximal tenderness. Subjects will apply a single patch at home approximately every 12 hours (e.g., morning and evening patch applications) for 14 days. Subjects will remove each patch after 4 hours. Subjects will have the option of applying the Synera patch as needed for an additional 2 week period (weeks 2-4) if they feel their shoulder impingement pain is severe enough to warrant treatment. Patches will be applied every 12 hours for up to 4 hours as needed during this period.
  Interventions: Drug: Synera® (lidocaine 70 mg and tetracaine 70 mg) topical patch
- Subacromial Injection (Active Comparator): A single injection will be administered into the subacromial space utilizing triamcinolone acetonide at the baseline visit.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Synera® (lidocaine 70 mg and tetracaine 70 mg) topical patch — Synera consists of a thin, uniform layer of a local anesthetic formulation with an integrated, oxygen-activated heating component that is intended to enhance the delivery of the local anesthetics. The drug formulation is an emulsion in which the oil phase is a eutectic mixture of lidocaine 70 mg and tetracaine 70 mg. The surface area of the entire Synera patch is approximately 50 cm2, 10 cm2 of which is active. The 40 cm2 perimeter is a medical grade adhesive. The Synera patches used in this study are the commercially available form.
  Other Names: lidocaine 70 mg/tetracaine 70mg topical patch
  Arms: Patch
Drug: Triamcinolone Acetonide — Triamcinolone Acetonide is a synthetic glucocorticoid corticosteroid with marked anti-inflammatory action, in a sterile aqueous suspension suitable for intralesional and intra-articular injection. Each mL of the sterile aqueous suspension provides 40 mg of triamcinolone acetonide, with sodium chloride for isotonicity, 0.9% (w/v) benzyl alcohol as a preservative, 0.75% carboxymethylcellulose sodium, and a 0.04% polysorbate 80; sodium hydroxide or hydrochloric acid may have been added to adjust pH between 5.0 and 7.5. At the time of manufacture, the air in the container is replaced by nitrogen.
  Other Names: Kenalog; Trivaris
  Arms: Subacromial Injection

SUMMARY:
Objective:

This purpose of this pilot study is to explore the potential usefulness of Synera for the treatment of pain associated with shoulder impingement syndrome.

DETAILED DESCRIPTION:
Subjects will receive either a subacromial injection at baseline or will be issued Synera patches to use daily for 2 weeks and then PRN for an additional 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age.
* have pain associated with shoulder impingement syndrome in a single shoulder (minimum 2-week duration).
* have tenderness at the attachment site of the rotator cuff tendons.
* have positive Hawkin's and Neer's signs.
* report an average pain intensity score of 4 (on an 11-point scale) over the past 24 hours at the Screening/Baseline visit.

Exclusion Criteria:

* have used any topically applied pain medication on the target treatment area within 14 days preceding Study Day 1, such as non-steroidal anti-inflammatory drugs (NSAIDs), menthol, methyl salicylate, local anesthetics (including Lidoderm®), or steroids.
* have used any injected medication within 60 days preceding Study Day 1, such as local anesthetic (lidocaine) or steroids.
* have a clinically significant illness within 14 days of Screening/Day 1 that, in the opinion of the investigator, would preclude the subject from participating in the study.
* are receiving class 1 antiarrhythmic drugs (ie, tocainide, mexiletine, etc.)
* have a history of and/or past diagnosis of severe hepatic disease.
* have participated in a clinical trial of an unapproved drug within 30 days prior to screening.
* are pregnant, breastfeeding, or a female of childbearing potential and not practicing an acceptable method of birth control.
* are unable or unwilling, in the opinion of the investigators, to comply with all study procedures and cooperate fully with research staff.
* have filed a disability claim or are currently receiving disability payments for shoulder impingement syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 6 weeks
  Average pain and worst pain over past 24 hours will be measured.

SECONDARY OUTCOMES:
Patient Global Assessment of Treatment Satisfaction | 6 weeks
Patient Global Impression of Change | 6 weeks
Pain Interference | 6 weeks
  Pain interference as it relates to general activity, normal work, and sleep will be measured at each visit.
Patch Site Evaluation for Erythema | 6 weeks
  site patch is applied will be assessed for erythema and patch site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Radnovich, DO, Principal Investigator — Injury Care Medical Center
Locations (1):
- Injury Care Medical Center, Boise, Idaho, United States